CLINICAL TRIAL: NCT03479138
Title: Non-Eosinophilic Neutrophilic Asthma
Acronym: ANNE
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Spanish Clinical Research Network - SCReN (Network)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ANN-2017-77
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2022-10

CONDITIONS: Neutrophilic Asthma
Keywords: severe asthma; induced sputum; asthma phenotypes; neutrophilic inflammation; microbiome
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Induced Sputum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neutrophilic asthma: Patients 18 to 80 years old diagnosed of severe asthma, requiring treatment at least with long acting beta agonists (LABA) + high doses inhaled corticosteroids (ICS) with eosinophil count in blood<300/mm3. They must be ex-smokers with less than 10 packs-year and no other relevant pulmonary disease.
  Interventions: Diagnostic Test: Induced sputum
- Non neutrophilic asthma: Patients 18 to 80 years old diagnosed of severe asthma, requiring treatment at least with LABA+ high doses ICS, with eosinophil count in blood<300/mm3. They must be ex-smokers with less than 10 packs-year and no other relevant pulmonary disease.
  Interventions: Diagnostic Test: Induced sputum

INTERVENTIONS:
Diagnostic Test: Induced sputum — Characterization with flow cytometry of the phenotype of the neutrophils isolated in the sputum, microbiome

SUMMARY:
Define and characterize the neutrophilic phenotype of severe asthma.

DETAILED DESCRIPTION:
Neutrophilic asthma (NA) is the asthma phenotype less known, causes a severe disease and does not have a specific treatment. Research on the neutrophilia mechanisms, new neutrophil (NEU) types and bronchial microbiome, can provide an opportunity to better understand the NA pathogenesis.

OBJECTIVES: 1. To describe the clinical characteristics of NA and its sub-phenotypes (SUBSTUDY 1); 2. To determine the NEU types associated with the NA and its sub-phenotypes (SUBSTUDY 2); and 3. To identify the bronchial microbiological flora of the NA, specifically related to lung microbiome and the immune response against Chlamydia Pneumoniae (SUBSTUDY 3).

METHODS: Multicenter prospective study including 100 patients with severe asthma (GINA/GEMA criteria): 50 with non-neutrophilic asthma (<65% NEU in induced sputum [IS]); and 50 with NA (> 64% NEU in IS). SUBSTUDY 1: clinical variables (years of evolution, exacerbations, asthma control test, mini asthma quality of life questionnary), comorbidities (GERD, nasal polyposis, obesity, ASS), pulmonary function (FEV1, exhaled fraction of nitric oxide, total lung capacity, Aspergillus), prick-test and CT scan chest; SUBSTUDY 2 (in IS and plasma): apoptotic index by means NE culture and flux cytometer (Annexin-V-FITC), NEU phenotype by surface markers (CD16, CD66b, CD62L, HLADR, CD177, CD11b, CD63, CXCR2, CXCR4) with density gradient study and determination of cytokines (IL-6, IL-8, IL-17, IL-1, IL-22) by ELISA; SUBSTUDY 3 (in IS): bronchial microbiome for 16 subunit rRNA by Phylogenetic Investigation of Communities by Reconstruction of Unobserved States (PICRUSt), and anti-Chlamydia Pneumoniae Immunoglobuling A by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years old
* Confirmed diagnosis of asthma (according to spanish guideline GEMA)
* Severe persistent asthma (step 5-6 GEMA)
* Eosinophils<300/mm3 in peripheral blood

Exclusion Criteria:

* Respiratory infection during the previous month
* Significant lung pathology not attributable to asthma (bronchiectasis with Reiff score>3)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients bewteen 18-80 years with severe asthma.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Phenotype of neutrophils | 24 hours
  To determine the types of neutrophils (in induced sputum and blood) associated with neutrophilic asthma and its subphenotypes according to flow cytometry
Microbiome analysis | 6 months
  To analyse the bronchial microbiological flora of neutrophilic asthma

SECONDARY OUTCOMES:
Clinical demographic characteristics | 1 year
  To describe the clinical characteristics and natural history of the neutrophilic asthma and its subphenotypes
Demographic characteristics | 1 year
  To describe demographic characteristics

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau. Carrer Mas Casanovas 90., Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nair P, Aziz-Ur-Rehman A, Radford K. Therapeutic implications of 'neutrophilic asthma'. Curr Opin Pulm Med. 2015 Jan;21(1):33-8. doi: 10.1097/MCP.0000000000000120. PMID 25415406
- [Background] Wenzel SE, Szefler SJ, Leung DY, Sloan SI, Rex MD, Martin RJ. Bronchoscopic evaluation of severe asthma. Persistent inflammation associated with high dose glucocorticoids. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):737-43. doi: 10.1164/ajrccm.156.3.9610046. PMID 9309987
- [Background] Simpson JL, Baines KJ, Ryan N, Gibson PG. Neutrophilic asthma is characterised by increased rhinosinusitis with sleep disturbance and GERD. Asian Pac J Allergy Immunol. 2014 Mar;32(1):66-74. doi: 10.12932/AP0322.32.1.2014. PMID 24641293
- [Background] Shaw DE, Berry MA, Hargadon B, McKenna S, Shelley MJ, Green RH, Brightling CE, Wardlaw AJ, Pavord ID. Association between neutrophilic airway inflammation and airflow limitation in adults with asthma. Chest. 2007 Dec;132(6):1871-5. doi: 10.1378/chest.07-1047. Epub 2007 Oct 9. PMID 17925424
- [Background] Wenzel SE. Asthma phenotypes: the evolution from clinical to molecular approaches. Nat Med. 2012 May 4;18(5):716-25. doi: 10.1038/nm.2678. PMID 22561835
- [Background] Simpson JL, Powell H, Boyle MJ, Scott RJ, Gibson PG. Clarithromycin targets neutrophilic airway inflammation in refractory asthma. Am J Respir Crit Care Med. 2008 Jan 15;177(2):148-55. doi: 10.1164/rccm.200707-1134OC. Epub 2007 Oct 18. PMID 17947611
- [Background] Polosa R, Thomson NC. Smoking and asthma: dangerous liaisons. Eur Respir J. 2013 Mar;41(3):716-26. doi: 10.1183/09031936.00073312. Epub 2012 Aug 16. PMID 22903959
- [Background] Sutherland ER, Martin RJ. Asthma and atypical bacterial infection. Chest. 2007 Dec;132(6):1962-6. doi: 10.1378/chest.06-2415. PMID 18079229
- [Background] Uddin M, Nong G, Ward J, Seumois G, Prince LR, Wilson SJ, Cornelius V, Dent G, Djukanovic R. Prosurvival activity for airway neutrophils in severe asthma. Thorax. 2010 Aug;65(8):684-9. doi: 10.1136/thx.2009.120741. PMID 20685741
- [Background] Newcomb DC, Peebles RS Jr. Th17-mediated inflammation in asthma. Curr Opin Immunol. 2013 Dec;25(6):755-60. doi: 10.1016/j.coi.2013.08.002. Epub 2013 Sep 11. PMID 24035139
- [Background] Chesne J, Braza F, Mahay G, Brouard S, Aronica M, Magnan A. IL-17 in severe asthma. Where do we stand? Am J Respir Crit Care Med. 2014 Nov 15;190(10):1094-101. doi: 10.1164/rccm.201405-0859PP. PMID 25162311
- [Background] Bruijnzeel PL, Uddin M, Koenderman L. Targeting neutrophilic inflammation in severe neutrophilic asthma: can we target the disease-relevant neutrophil phenotype? J Leukoc Biol. 2015 Oct;98(4):549-56. doi: 10.1189/jlb.3VMR1214-600RR. Epub 2015 May 14. PMID 25977288
- [Background] Pillay J, Ramakers BP, Kamp VM, Loi AL, Lam SW, Hietbrink F, Leenen LP, Tool AT, Pickkers P, Koenderman L. Functional heterogeneity and differential priming of circulating neutrophils in human experimental endotoxemia. J Leukoc Biol. 2010 Jul;88(1):211-20. doi: 10.1189/jlb.1209793. Epub 2010 Apr 16. PMID 20400675
- [Background] Beyrau M, Bodkin JV, Nourshargh S. Neutrophil heterogeneity in health and disease: a revitalized avenue in inflammation and immunity. Open Biol. 2012 Nov;2(11):120134. doi: 10.1098/rsob.120134. PMID 23226600
- [Background] Green BJ, Wiriyachaiporn S, Grainge C, Rogers GB, Kehagia V, Lau L, Carroll MP, Bruce KD, Howarth PH. Potentially pathogenic airway bacteria and neutrophilic inflammation in treatment resistant severe asthma. PLoS One. 2014 Jun 23;9(6):e100645. doi: 10.1371/journal.pone.0100645. eCollection 2014. PMID 24955983
- [Background] Kiley JP, Caler EV. The lung microbiome. A new frontier in pulmonary medicine. Ann Am Thorac Soc. 2014 Jan;11 Suppl 1(Suppl 1):S66-70. doi: 10.1513/AnnalsATS.201308-285MG. No abstract available. PMID 24437410
- [Background] Marri PR, Stern DA, Wright AL, Billheimer D, Martinez FD. Asthma-associated differences in microbial composition of induced sputum. J Allergy Clin Immunol. 2013 Feb;131(2):346-52.e1-3. doi: 10.1016/j.jaci.2012.11.013. Epub 2012 Dec 23. PMID 23265859
- [Background] Huang YJ, Nariya S, Harris JM, Lynch SV, Choy DF, Arron JR, Boushey H. The airway microbiome in patients with severe asthma: Associations with disease features and severity. J Allergy Clin Immunol. 2015 Oct;136(4):874-84. doi: 10.1016/j.jaci.2015.05.044. Epub 2015 Jul 26. PMID 26220531
- [Background] Martin RJ, Kraft M, Chu HW, Berns EA, Cassell GH. A link between chronic asthma and chronic infection. J Allergy Clin Immunol. 2001 Apr;107(4):595-601. doi: 10.1067/mai.2001.113563. PMID 11295645
- [Background] Brusselle GG, Vanderstichele C, Jordens P, Deman R, Slabbynck H, Ringoet V, Verleden G, Demedts IK, Verhamme K, Delporte A, Demeyere B, Claeys G, Boelens J, Padalko E, Verschakelen J, Van Maele G, Deschepper E, Joos GF. Azithromycin for prevention of exacerbations in severe asthma (AZISAST): a multicentre randomised double-blind placebo-controlled trial. Thorax. 2013 Apr;68(4):322-9. doi: 10.1136/thoraxjnl-2012-202698. Epub 2013 Jan 3. PMID 23291349
- [Background] Blasi F. Atypical pathogens and respiratory tract infections. Eur Respir J. 2004 Jul;24(1):171-81. doi: 10.1183/09031936.04.00135703. PMID 15293621
- [Background] Frehn L, Jansen A, Bennek E, Mandic AD, Temizel I, Tischendorf S, Verdier J, Tacke F, Streetz K, Trautwein C, Sellge G. Distinct patterns of IgG and IgA against food and microbial antigens in serum and feces of patients with inflammatory bowel diseases. PLoS One. 2014 Sep 12;9(9):e106750. doi: 10.1371/journal.pone.0106750. eCollection 2014. PMID 25215528
- [Background] Tuuminen T, Edelstein I, Punin A, Kislova N, Stratchounski L. Use of quantitative and objective enzyme immunoassays to investigate the possible association between Chlamydia pneumoniae and Mycoplasma pneumoniae antibodies and asthma. Clin Microbiol Infect. 2004 Apr;10(4):345-8. doi: 10.1111/j.1198-743X.2004.00822.x. PMID 15059128
- See also: Website of the spanish guideline of asthma — https://www.gemasma.com/
- See also: Website of the european guideline of asthma — http://ginasthma.org/